CLINICAL TRIAL: NCT06325280
Title: Utilizing Exercise Cardiovascular and Skeletal Magnetic Resonance Imaging to Evaluate Factors Associated With Cardiorespiratory Fitness in Children With Acquired and Congenital Heart Disease
Brief Title: Exercise MRI to Evaluate Cardiorespiratory Fitness in Children With Heart Disease
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00132542
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pediatric ALL; Congenital Heart Disease; Heart Transplantation
Keywords: Pediatric cardiology; Exercise cardiac MRI
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Heart Defects, Congenital | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital heart disease: Participants aged 10-18 years who have congenital heart disease.
  Interventions: Diagnostic Test: Exercise cardiac MRI Assessment; Diagnostic Test: Cardiopulmonary Exercise Test
- Heart transplant recipient: Participants aged 10-18 years who have recieved a heart transplant.
  Interventions: Diagnostic Test: Exercise cardiac MRI Assessment; Diagnostic Test: Cardiopulmonary Exercise Test

INTERVENTIONS:
Diagnostic Test: Exercise cardiac MRI Assessment — Participants will undergo a standard cardiac MRI to assess resting ventricular structure and function then complete an exercise cardiac MRI assessment using an MRI-compatible stepping ergometer.
Diagnostic Test: Cardiopulmonary Exercise Test — Cardiopulmonary exercise testing will be performed using a cycle ergometer. Consistent with standard guidelines, workload will progressively increase (10W ramp protocol) such that peak oxygen consumption (VO2peak) is achieved within 8-12 minutes. VO2peak, VO2 at anaerobic threshold, peak power output (PPO), ventilation/carbon dioxide production (VE/VCO2) slope, peak heart rate (HR), and HR recovery at 1- and 3-minutes will be recorded. VO2peak will be converted to age-, weight, and sex-specific norms and a %predicted value.
  Other Names: CPET

SUMMARY:
There are many barriers to heart-healthy lifestyles in pediatric patients with acquired and congenital heart disease. Investigators want to further understand how participants heart and skeletal muscles work together during exercise and evaluate the impact on cardiac function. To do this, the investigators will use magnetic resonance imaging (MRI) to scan the heart and skeletal muscles during exercises to assess blood flow, oxygenation and function.

DETAILED DESCRIPTION:
Exercise cardiac MRI's are the non-invasive gold standard for assessing biventricular function during exercise. While exercise MRI has not been previously studied in pediatric HTRs, it has been effectively utilized in children with single ventricle congenital heart disease. The purpose of this study is to fully understand the cardiac adaptations induced by exercise training.

Primary objective: Evaluate the association between exercise MRI cardiac and skeletal muscle measures and cardiorespiratory fitness in pediatric acquired (HTRx) and CHD participants.

Hypothesis: Cardiac adaptations to exercise and skeletal muscle functioning will be positively associated with measured CRF in CHD patients and those post-transplant.

Secondary objective: Evaluate changes in exercise MRI measures of cardiac and skeletal muscle function following a 12-week high-intensity interval training (HIIT) exercise protocol in children with acquired and congenital heart disease.

Hypothesis: a 12-week HIIT intervention will result in improvements in cardiac and skeletal muscle responses to exercise.

This will be a single-center, prospective observational study.

Participants will include 10-18 year old pediatric heart transplant recipients (HTR) and congenital heart disease (CHD) patients followed at the Stollery Children's Hospital.

Participants will undergo cardiopulmonary exercise testing (CPET) using a cycle ergometer and standardized protocols. On a separate day (within 2 weeks of the testing), participants will return and undergo a standard cardiac MRI to assess resting ventricular structure and function. They will then complete an exercise cardiac MRI assessment using an MRI-compatible stepping ergometer.

Participants and their parent will also be asked to complete questionnaires to determine their feelings towards exercise and physical activity.

As this will be a single-center study. The analysis will be largely exploratory and the sample size will be determined based on the available patient population. Based on a review of potentially eligible participants at our center, the investigators anticipate recruiting 10 participants post-HTR and 10 CHD participants to evaluate the primary objective. As the secondary objective (changes in cardiac and skeletal muscle MRI measures) requires repeated assessments and involvement in the MedBIKE™ HIIT trial, recruitment to address this objective may be lessened; the investigators thus anticipate recruiting ~6 participants post-transplant and 6 participants with CHD. The statistical analysis will be carried out in collaboration with the Women and Children's Health Research Institute (WCHRI) biostatistics team (accounted for in budget). Differences in MRI and CPET measures among participants, and changes in the measures (Objective 2) will be evaluated by independent t-tests or Mann-Whitney tests for continuous variables and chi-square or Fisher's exact tests for categorical variables. Pearson correlations will be used to evaluate associations between VO2peak (and other CPET measures of CRF) and measures of cardiac function and output and peripheral muscle oxygen extraction.

ELIGIBILITY:
Inclusion Criteria:

* 10 - 18 year olds followed at the Stollery Children's Hospital
* Heart transplant recipients ≥6 months post-transplant
* Have a moderate-complex congenital heart disease diagnosis

Exclusion Criteria:

* Non-English speaking
* Exercise restricted by the patient's clinical cardiologist
* Clinical antibody- or cellular-mediated rejection within 3-months of the assessment or during the study period (for HTRs)
* Previous involvement in a CR or exercise intervention program
* Previous exercise stress test demonstrating sustained arrhythmias, ST segment elevation or depression greater than 3mm, an inappropriate rise in blood pressure (BP) (<20 mmHg) or a systolic BP >200 mmHg, or symptoms of chest pain or syncope
* Resting arterial saturation <85% or oxygen requirements
* Moderate ventricular systolic dysfunction (or worse) at the most recent echocardiogram
* History of chest pain on exertion; unrepaired/unpalliated CHD
* Arrhythmias in the last year (including supraventricular tachycardia, ventricular tachycardia, atrioventricular block or history of (Mobitz II or worse))
* New York Heart Association class II or worse symptoms
* Active medical inter-current illness limiting ability to participate
* Cognitive impairment limiting the communication needed for the exercise MRI
* Research MRI contraindications (e.g. any type of pacemaker), or any orthopedic limitation preventing exercise testing
* Extracardiac or congenital abnormality limiting the participant's functional ability to exercise
* Pregnant

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants in this study will be 10-18 year olds, with acquired or congenital heart disease, that are followed by the Stollery Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI assessment of cardiac structure at rest | Baseline
  Participants will undergo a standard cardiac MRI using a Siemens MAGNETOM Prisma 3.0T CMR (Siemens Healthineers, Erlangen, Germany) for the assessment of resting ventricular structure.
MRI assessment of cardiac function at rest | Baseline
  Participants will undergo a standard cardiac MRI using a Siemens MAGNETOM Prisma 3.0T CMR (Siemens Healthineers, Erlangen, Germany) for the assessment of resting ventricular function.
Maximal exercise MRI assessment of cardiac structure | Baseline
  Participants will undergo an exercise cardiac MRI assessment using an MRI-compatible stepping ergometer (Cardio Step Module, Ergospect) to assess cardiac output.
Cardioplumonary Exercise Test | Baseline
  Participants will undergo a cardiopulmonary exercise test using a cycle ergometer to assess VO2peak.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Khoury, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. All data will be de-identified prior to analysis and published.

REFERENCES:
- [Background] Khoury M, Phillips DB, Wood PW, Mott WR, Stickland MK, Boulanger P, Rempel GR, Conway J, Mackie AS, Khoo NS. Cardiac rehabilitation in the paediatric Fontan population: development of a home-based high-intensity interval training programme. Cardiol Young. 2020 Oct;30(10):1409-1416. doi: 10.1017/S1047951120002097. Epub 2020 Jul 27. PMID 32716280
- [Background] Spence C, Khoo N, Mackie A, Conway J, Rowland S, Foshaug R, Boulanger P, Spence JC, Stickland MK, Khoury M. Exploring the Promise of Telemedicine Exercise Interventions in Children and Adolescents With Congenital Heart Disease. Can J Cardiol. 2023 Nov;39(11S):S346-S358. doi: 10.1016/j.cjca.2023.08.015. Epub 2023 Aug 30. PMID 37657493
- [Background] Spence CM, Foshaug R, Rowland S, Krysler A, Conway J, Urschel S, West L, Stickland M, Boulanger P, Spence JC, Khoury M. Evaluating a Telemedicine Video Game-Linked High-Intensity Interval Training Exercise Programme in Paediatric Heart Transplant Recipients. CJC Pediatr Congenit Heart Dis. 2023 Apr 11;2(4):198-205. doi: 10.1016/j.cjcpc.2023.04.001. eCollection 2023 Aug. PMID 37969861